CLINICAL TRIAL: NCT06911931
Title: Visual Perception in Schizophrenia: Assessing Predictive Processing in the Earliest Stages of the Visual Cortical Hierarchy
Brief Title: Visual Perception in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Edmund Lalor, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00007500; R21MH140245 (NIH)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia Disorders; Bipolar Disorder; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental)
  Interventions: Other: EEG measure of visual processing

INTERVENTIONS:
Other: EEG measure of visual processing — Non-invasive scalp EEG measure of early cortical visual processing.

SUMMARY:
This study aims to identify novel markers of psychosis using electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

* All Subjects
* Aged 18-65
* 20/32 visual acuity or better (using in-house optical correction, if necessary)
* An ability to speak English well enough to complete study assessments and to consent to the study
* Subjects with Schizophrenia-Spectrum Disorder
* Meets DSM-5 diagnostic criteria for schizophrenia, schizoaffective disorder, or schizophreniform disorder as confirmed by the Structured Interview for DSM-5 (SCID-5).
* Subjects with Bipolar Disorder
* Meets DSM-5 diagnostic criteria for bipolar disorder (type I, II, or unspecified) as confirmed by the Structured Interview for DSM-5 (SCID-5).

Exclusion Criteria:

* All subjects
* Presence of characteristics that could impair one's ability to comprehend the nature of the study, provide informed consent, or understand the assessment questions, including the following:

  * Subject cannot read and understand the instructions well enough to complete the tasks or cannot provide informed consent.
  * Intellectual impairment (WRAT-5 score < 70) (at the discretion of experimenter);
  * Actively intoxicated, as shown via patient self-report or staff report;
  * Substance use disorder in the past 3 months;
  * Subject considered high risk for suicidal acts (i.e., active suicidal ideation as determined by clinical interview OR any suicide attempt in 30 days prior to screening);
  * Subject violence (involving severe/lethal means or violence occurring in prior 6 months) or extreme agitation.
  * Being in a current manic state
  * Head injury with loss of consciousness greater than 10 minutes (at the discretion of the experimenter).
  * Subject has had electroconvulsive therapy (ECT) in the past 8 weeks;
  * Diagnosed with a neurological condition (tumor, stroke, brain injury) or neurological disorder, including seizure disorders. Diagnosed with pervasive developmental disorder (phone screen or medical records)
  * Lazy eye or squint or other known ocular pathology
* Healthy Control Subjects
* Any lifetime psychotic disorder or history of psychiatric hospitalization (self disclosure);
* Daily antidepressant, mood stabilizer or antipsychotic medication use in the last 6 months, or benzodiazepine use during the prior 2 days (self-disclosure); iii. First-degree relative(s) with a schizophrenia spectrum disorder (based on subject self-report) or bipolar disorder.
* Case-match Control Non-ill Subjects
* Any lifetime psychotic disorder (as assessed by SCID/or SSD);
* Recurrent depressive episodes or being in a current depressive episode (as assessed by SCID/or SSD)
* Persistent threshold psychotic symptoms
* History of psychiatric hospitalization;
* Daily antidepressant, mood stabilizer or antipsychotic medication use in the last 6 months, or benzodiazepine use during the prior 2 days
* First-degree relative(s) with a schizophrenia spectrum disorder (based on subject self-report) or bipolar disorder.
* Bipolar Subjects
* Persistent threshold psychotic symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
mean amplitude of EEG visual response | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes